CLINICAL TRIAL: NCT06138015
Title: Effect of Time-restricted Eating on Cognitive Function and Other Biopsychosocial Factors in Menopausal Women Undertaking a 12-week Exercise Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BJozwiak_PhD
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Menopause; Cognitive Deficits, Mild
MeSH Terms: conditions — Cognition Disorders; Lymphoma, Follicular | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and Time-Restricted Eating (Experimental)
  Interventions: Behavioral: Exercise and Time-Restricted Eating
- Exercise only (Active Comparator)
  Interventions: Behavioral: Exercise only

INTERVENTIONS:
Behavioral: Exercise and Time-Restricted Eating — Moderate intensity circuit mixed endurance and resistance exercise programme two times per week for 55 minutes for 12 weeks and a time-restricted eating following 16:8 protocol for 12 weeks.
  Arms: Exercise and Time-Restricted Eating
Behavioral: Exercise only — Moderate intensity circuit mixed endurance and resistance exercise programme two times per week for 55 minutes for 12 weeks only.
  Arms: Exercise only

SUMMARY:
The goal of this quasi-experimental study is to test effect of time-restricted eating on cognitive function and other biopsychosocial factors in menopausal women undertaking a 12-week exercise programme. The main questions to answer are:

1. What is effect of time-restricted eating on cognitive function in menopausal women undertaking a 12-week exercise programme?
2. What is effect of time-restricted eating on menopausal symptoms in menopausal women undertaking a 12-weeks exercise programme?
3. What is effect of time-restricted eating on metabolic health parameters in menopausal women undertaking a 12-weeks exercise programme?

Participants of both groups will have moderate intensity circuit mixed endurance and resistance exercise programme two times per week for 55 minutes for 12 weeks. Participants of one of two groups will not only exercise but also have a time-restricted eating following 16:8 protocol for 12 weeks.

Participants will have pre-tests and post-tests:

* blood samples collection (to measure level of brain-derived neurotrophic factor, glial cell derived neurotrophic factor, insulin, glucose, lipid profile),
* body composition analysis,
* Stroop test and N-back test,
* electroencephalography using Emotiv Epic X devices,
* One-repetition maximum test, Ruffier test,
* Questionnaire assessment (using Menopause Rating Scale and The Menopause-Specific Quality of Life Questionnaire).

Researchers will compare two groups - exercise group and combination group which will do both time-restricted eating and exercise to see if there is a modulating effect of time-restricted eating in participants undertaking exercise.

ELIGIBILITY:
Inclusion Criteria:

* perimenopause, menopause or post-menopause
* lightly physically active or physically inactive

Exclusion Criteria:

* using hormone replacement therapy or hormonal contraception
* having significant contraindications to physical exercise or time-restricted eating

Ages: 41 Years to 61 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Brain-derived neurotrophic factor | Before and after 12-week intervention
  Level of brain-derived neurotrophic factor in ng/ml
Glial cell derived neurotrophic factor | Before and after 12-week intervention
  Level of glial cell derived neurotrophic factor in ng/ml
Insulin | Before and after 12-week intervention
  Level of insulin in μIU/ml
Glucose | Before and after 12-week intervention
  Level of glucose in mg/dl
LDL-cholesterol | Before and after 12-week intervention
  Level of cholesterol LDL in mg/dl
Muscle mass | Before and after 12-week intervention
  Bioelectrical impedance analysis for estimating body composition, in particular muscle mass in kg
Fat mass | Before and after 12-week intervention
  Bioelectrical impedance analysis for estimating body composition, in particular fat mass in kg
Stroop test | Before and after 12-week intervention
  Cognitive functions assessment with Stroop test in points. Higher scores means better outcome.
N-back test | Before and after 12-week intervention
  Cognitive functions assessment with N-back test in points. Higher scores means better outcome.
Electroencephalography | Before and after 12-week intervention
  Measurement of brain waves (alpha, beta, gamma, theta) to assess electrical activity of the brain using Emotiv Epoc X device
One-repetition maximum test | Before and after 12-week intervention
  Strength assessment with one-repetition maximum test in kg
Ruffier test | Before and after 12-week intervention
  Cardiorespiratory fitness assessment with Ruffier test in points. Minimum value is 0, maximum value is 10. Higher score means worse outcome.
Menopause Rating Scale | Before and after 12-week intervention
  Menopausal symptoms assessment with Menopause Rating Scale in points. Minimum value is 0 and maximum value is 44. Higher score means worse outcome.
The Menopause-Specific Quality of Life Questionnaire | Before and after 12-week intervention
  Menopausal symptoms assessment with The Menopause-Specific Quality of Life Questionnaire in points. Minimum value is 0 and maximum value is 174. Higher score means worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Physical Education, Poznan, Greater Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jozwiak B, Kleka P, Laudanska-Krzeminska I. Effect of exercise alone and in combination with time-restricted eating on cognitive health in menopausal women. Front Public Health. 2025 Aug 13;13:1640512. doi: 10.3389/fpubh.2025.1640512. eCollection 2025. PMID 40880914
- [Derived] Jozwiak B, Domin R, Krzywicka M, Laudanska-Krzeminska I. Effect of exercise alone and in combination with time-restricted eating on cardiometabolic health in menopausal women. J Transl Med. 2024 Oct 21;22(1):957. doi: 10.1186/s12967-024-05738-y. PMID 39434160